CLINICAL TRIAL: NCT06157177
Title: Efficacy of Modified Release Metaxalone 640 mg in Acute Lumbosacral Musculoskeletal Conditions With Spinal Stenosis and Sciatica
Brief Title: Efficacy of M640 in Acute Lumbosacral Musculoskeletal Conditions.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Illumination Health (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMMSS-01
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Sciatica Acute; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — metaxalone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active M640 (Active Comparator): Metaxalone micronized 640 mg over encapsulated tablet Taken orally every 6 hours for 7 days
  Interventions: Drug: Metaxalone 640 mg Oral Tablet
- Placebo (Placebo Comparator): Inactive placebo capsule 640 mg Taken orally every 6 hours for 7 days
  Interventions: Drug: Metaxalone 640 mg Oral Tablet

INTERVENTIONS:
Drug: Metaxalone 640 mg Oral Tablet — Metaxalone 640 mg used for the treatment of discomforts associated with acute, musculoskeletal pain.
  Other Names: Skelaxin un-micronized; M640; metaxalone micronized

SUMMARY:
The goal of this clinical trial is to learn if a modification to metaxalone 640 mg can reduce low back and leg pain. The participants will be 18 to 80 years old, healthy with newly occurring back or leg pain. The main question aims to compare a group taking active treatment and a group taking a look-alike substance containing no active treatment. All participants will answer questions on Day 1, before treatment, and on 7-day after treatment, about:

* Amount and quality of pain
* Interference with physical activity
* Interference with sleep

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled, multi-center study of metaxalone 640 mg plus standard of care for patients with acute lumbo sacral musculoskeletal conditions with spinal stenosis and sciatica. Participants will be randomized 1:1. Following the initial pilot-study a second study will randomize a larger population of patients with appropriate power.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant conditions impacting quality or quantity of pain
* Baseline Numeric Pain Scale ≥ 6
* Capable of answering text or email survey reminders
* Low back pain with or without sciatica

Exclusion Criteria:

* Current use of other skeletal relaxants
* Current use of other pain relievers
* Current use of cimetidine or monoamine oxidase inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change of Numeric Pain Scale | Day 1 to Day 7
  Change from Baseline in low back pain and leg pain as measured by the Numeric Pain Rating Scale (NPRS) at Day 7

CONTACTS AND LOCATIONS:
Overall Officials: S Sodhi, Study Director — Illumination Health
Locations (19):
- United States (19):
  - East Alabama Arthritis Center, Auburn, Alabama
  - Sean Wollaston, MD, Valley Village, California
  - Arthritis and Osteoporosis Center, Aventura, Florida
  - William Sunshine, MD, Boca Raton, Florida
  - Robert Levin, MD, Clearwater, Florida
  - 5. CZ Rheumatology, Coral Springs, Florida
  - 4. Palm Beach Rheumatology and Wellness, Jupiter, Florida
  - Family Arthritis Center, Loxahatchee Groves, Florida
  - Arthritis and Rheumatology Center of South Florida, Margate, Florida
  - Arthritis and Rheumatic Care Center, South Miami, Florida
  - Arthritis Research and Treatment Center, Stockbridge, Georgia
  - Jayashree Sinha, MD 1, Clovis, New Mexico
  - Carolina Rheumatology, Fayetteville, North Carolina
  - Ohio Arthritis and Osteoporosis Center of Southwest Ohio, Springboro, Ohio
  - Heritage Rheumatology & Arthritis Care, Colleyville, Texas
  - Integrative Rheumatology of South Texas, Harlingen, Texas
  - Southwest Research Group, Mesquite, Texas
  - DFW Rheumatology, Red Oak, Texas
  - Northern Virginia Center for Arthritis, Annandale, Virginia

IPD SHARING:
Plan to Share IPD: No